CLINICAL TRIAL: NCT04135014
Title: Intranasal Dexmedetomidine or Oral Midazolam Alone Versus Combination With Intranasal Dexmedetomidine and Oral Midazolam for Premedication in Pediatric Patients Undergoing Minor Surgery
Brief Title: Combination With Intranasal Dexmedetomidine and Oral Midazolam for Premedication in Pediatric Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2019-03-111
Record Dates: First submitted 2019-10-17; First posted 2019-10-22 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Midazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Midazolam (Placebo Comparator): Patients were assigned to receive oral midazolam 0.5mg.kg-1 approximately 30-40 minutes before surgery using a computer-generated random number table.
  Interventions: Drug: Midazolam
- Dexmedetomidine (Experimental): Patients were assigned to receive intranasal dexmedetomidine 2ug/kg approximately 30-40 minutes before surgery using a computer-generated random number table.
  Interventions: Drug: Dexmedetomidine
- Midazolam and Dexmedetomidine (Experimental): Patients were assigned to receive intranasal dexmedetomidine 1ug.kg-1 and oral midazolam 0.5mg.kg-1 approximately 30-40 minutes before surgery using a computer-generated random number table.
  Interventions: Drug: Midazolam and Dexmedetomidine

INTERVENTIONS:
Drug: Midazolam — oral midazolam 0.5mg.kg-1 approximately 30-40 minutes before surgery using a computer-generated random number table.
  Other Names: oral midazolam
  Arms: Midazolam
Drug: Dexmedetomidine — intranasal dexmedetomidine 2µg.kg-1 approximately 30-40 mins before surgery using a computer-generated random number table.
  Other Names: intranasal dexmedetomidine
  Arms: Dexmedetomidine
Drug: Midazolam and Dexmedetomidine — oral midazolam 0.5mg.kg-1 and intranasal dexmedetomidine 1ug.kg-1 approximately 30-40 mins before surgery using a computer-generated random number table.
  Other Names: combination with intranasal dexmedetomidine and oral midazolam
  Arms: Midazolam and Dexmedetomidine

SUMMARY:
Children tend to anxiety and even fear before survey. And this kind of anxiety will not result in the forced induction of anesthesia, but also may increase the incidence of postoperative agitation in children, even lead to postoperative behavior changes.Currently,Oral midazolam or intranasal dexmedetomidine alone is commonly used as a preoperative regimen, but the clinical effects of each single-use are not satisfactory. In the investigators' study，the researchers conducted the current study to investigate whether dexmedetomidine combined with midazolam can increase the rate of satisfactory anesthesia induction in pediatric patients and achieve better sedative effect.

DETAILED DESCRIPTION:
A trained member of the research team obtained a baseline The Modified Yale Preoperative Anxiety Scale(mYPAS) after obtaining consent. And corresponding study medication is administered about 30-40 minutes before the anesthesia induction.Vital signs were measured every 5 min after study medication administration.The sedation scores of the children were recorded with University of Michigan Sedation Scale (UMSS) every 10 minutes.The onset time of satisfactory sedation and parental separation anxiety scale was noted.Then recorded the degree of cooperation during inhalation anesthesia induction and recovery times.Moreover, recorded the pediatric anesthesia emergence delirium scale (PAED) during the recovery period.

ELIGIBILITY:
Inclusion Criteria:

1. with American Society of Anesthesiologists (ASA) physical status I or II；
2. aged 2-6 years；
3. children with weight for age within the normal range
4. were scheduled lower abdominal and perineal surgery with an expected operation time shorter than 30 minutes.

Exclusion Criteria:

1. Children who had gastrointestinal,Cardiovascular or endocrine dysfunction;
2. contraindication to preoperative sedation or had a known allergy or hypersensitive reaction to either dexmedetomidine or midazolam;
3. with any nasal pathology,organ dysfunction;
4. recently respiratory infection, mental disorder;
5. other reasons that researchers hold it is not appropriate to participate in this trial.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 138 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
The degree of cooperation during inhalation anesthesia induction | During inhalation anesthesia induction
  Induction Compliance Checklist range from 0 through 10,and lower scores indicate the higher degree of cooperation during inhalation anesthesia induction

SECONDARY OUTCOMES:
Anxiety before induction of anesthesia | Before preoperative medication
  The Modified Yale Preoperative Anxiety Scale:
  The 22-item measure has five behavioural categories: activity, emotional expressivity, alertness and arousal, vocalizations, and interaction with parents. Total scores range from 23.33 through 100 with higher scores indicating greater anxiety.
The level of sedation | Each 10 minutes during the preoperative period
  University of Michigan Sedation Scale:
  0 -Awake/Alert
  1 -Minimally Sedated: Tired/sleepy, appropriate response to verbal conversation and/or sounds.
  2- Moderately Sedated: Somnolent/sleeping, easily aroused with light tactile stimulation.
  3 - Deeply Sedated: Deep sleep, arousable only with significant physical stimulation.
  4 - Unarousable.
  higher scores mean a higher levels of sedation.
The onset time of satisfactory sedation | During the preoperative period
  The onset time of satisfactory sedation, defined as the time from drug administration to the time when the University of Michigan Sedation Scale reached two points.
  University of Michigan Sedation Scale:
  0 -Awake/Alert
  1 -Minimally Sedated: Tired/sleepy, appropriate response to verbal conversation and/or sounds.
  2- Moderately Sedated: Somnolent/sleeping, easily aroused with light tactile stimulation.
  3 - Deeply Sedated: Deep sleep, arousable only with significant physical stimulation.
  4 - Unarousable.
  higher scores mean a higher levels of sedation.
Parental separation anxiety scale | During the preoperative period
  A four-point parental separation anxiety scale as follows:
  1. -Easy separation,
  2. -Whimpers, but is easily reassured, not clinging,
  3. - Cries and cannot be easily reassured, but not clinging to parents,
  4. - Crying and clinging to parents.
  The scores of 1 and 2 signified acceptable separation whereas scores of 3 and 4 were classified as difficult separation.
Recovery times | Within up to 30 minutes after child's first eye opening in the postoperative period
  The time from discontinuation of sevoflurane to the first open eye of the children and to achieve aldrete≥9
Pediatric anesthesia emergence delirium | Within up to 15-30 minutes after child's first eye opening in the postoperative period
  The pediatric anesthesia emergence delirium scale consists of four items. Each item is scored 0-4 yielding a total between 0 and 20.
  The degree of emergence delirium increased directly with the total score.pediatric anesthesia emergence delirium scale ≥12 at any time indicates presence of emergence delirium.
Number of children with adverse effects | Up to 24 hours including preoperative, intraoperative, and postoperative periods
  Number of children with adverse effects
  1. Bradycardia and/or hypotension need for hemodynamic support
  2. Desaturation is defined as Oxygen desaturation <90%
  3. Salivation
  4. Any adverse effects requiring interventions

CONTACTS AND LOCATIONS:
Overall Officials: Huacheng Liu, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University; Yuhang Cai, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No